CLINICAL TRIAL: NCT04866914
Title: Acceptance and Commitment Therapy for Chronic Insomnia in Adults
Brief Title: Acceptance and Commitment Therapy for Insomnia
Acronym: ACT-I
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 65743917.2.0000.0068
Record Dates: First submitted 2021-04-13; First posted 2021-04-30 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2021-05

CONDITIONS: Insomnia
Keywords: INSOMNIA; acceptance and commitment therapy; Cognitive behavioral therapy; SLEEP
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ACT for Insomnia (Experimental)
  Interventions: Behavioral: Acceptance and Commitment Therapy for Insomnia
- CBT for Insomnia (Active Comparator)
  Interventions: Behavioral: Cognitive Behavioral Therapy for Insomnia
- Wait List (No Intervention)

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy for Insomnia — ACT-I treatment group: Participants diagnosed with chronic insomnia will receive group treatment. The six sessions will be aimed at psychoeducation about sleep added to the therapeutic processes of acceptance, mindfulness, availability, values, defusion and commitment, used in ACT.
  Other Names: ACT-I
  Arms: ACT for Insomnia
Behavioral: Cognitive Behavioral Therapy for Insomnia — Active control group CBT-I: Participants diagnosed with chronic insomnia will receive treatment in a group. The six sessions will be aimed at cognitive-behavioral components, such as education and sleep hygiene, stimulus control, sleep restriction and demystification / restructuring of belief beliefs.
  Other Names: CBT-I
  Arms: CBT for Insomnia

SUMMARY:
Insomnia is a frequent complaint and is associated with impairments in physical and psychological health. Although Cognitive-Behavioral Therapy (CBT) demonstrates effective results for insomnia, there are those who do not respond to this type of intervention or present difficulties in adherence. Acceptance and Commitment Therapy (ACT) presents itself as a potentially useful intervention for the treatment of insomnia, for which, instead of focusing on controlling the symptoms, the respective approach focuses on accepting the feelings and thoughts associated, through value-based actions. The aim of this study is to evaluate the effectiveness of ACT for chronic insomnia in adults. Participants will be 150 adults aged between 18 and 59 years, diagnosed with chronic insomnia who will be randomly assigned to the ACT, CBT and wait list (WL) groups. For both groups (ACT and CBT), the intervention will be performed in six group and weekly sessions. Assessments of sleep patterns, insomnia, depression, anxiety, psychological flexibility, acceptance of sleep, beliefs about sleep, personality traits will be performed in the pre-treatment, post-treatment and six-month follow-up. After the intervention is completed, participants will respond to an inventory of compliance and satisfaction. Treatment effects will assessed using the fixed effects of group variables (ACT vs. CBT-I and ACT vs. waitlist) and their interaction with time (pre-test vs. post-test and pretest vs. six-month follow-up). Estimated pairwise contrasts to examine changes across time within groups will be used. Variables will analyzed using generalized mixed models (GMM).

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of chronic insomnia

Exclusion Criteria:

* Neurological degenerative disease
* Psychotic disorder
* sleep apnea, restless legs or periodic limb movements during sleep, or a circadian-based sleep disorder (e.g., delayed or advanced sleep phase syndrome)
* cognitive impairments
* unavailability in attending the sessions.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 227 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2023-03-15 (Actual); Study Completion 2023-03-15 (Actual)

PRIMARY OUTCOMES:
Change in the score of Insomnia Severity Index (ISI) | baseline, 7 weeks and 24 weeks after treatment commencement.
  Change in the total score of Insomnia Severity Index (ISI)

SECONDARY OUTCOMES:
Remission - categorical variable | baseline, 7 weeks and 24 weeks after treatment commencement.
  a final ISI score under 8 points
Treatment response - categorical variable | baseline, 7 weeks and 24 weeks after treatment commencement.
  change or reduction in the ISI total score of 8 points or more
Reduction in Sleep Onset Latency (SOL) | baseline, 7 weeks and 24 weeks after treatment commencement.
  Reduction in Sleep Onset Latency (SOL) measured by sleep diary
Reduction in Wake After Sleep Onset (WASO) | baseline, 7 weeks and 24 weeks after treatment commencement.
  Reduction in Wake After Sleep Onset (WASO) measured by sleep diary
Increase in Total Sleep Time (TST) | baseline, 7 weeks and 24 weeks after treatment commencement.
  Increase in Total Sleep Time (TST) measured by sleep diary
Increase in Sleep Efficiency (SE) | baseline, 7 weeks and 24 weeks after treatment commencement.
  Increase in Sleep Efficiency (SE) measured by sleep diary
Change in the Hospital Anxiety and Depression Scale (HADS) | baseline, 7 weeks and 24 weeks after treatment commencement.
  Change in the total score for the anxiety variable (HADAS-A) and total score for the depression variable (HADAS-D)
Change in the Acceptance and Action Questionnaire-II (AAQ-II) | baseline, 7 weeks and 24 weeks after treatment commencement.
  Change in the the total score of Acceptance and Action Questionnaire-II (AAQ-II)
Change in the Sleep Problem Acceptance Questionnaire (SPAQ) | baseline, 7 weeks and 24 weeks after treatment commencement.
  Change in the the total score of Sleep Problem Acceptance Questionnaire (SPAQ)
Change in the Dysfunctional Beliefs and Attitudes about Sleep (DBAS-16) | baseline, 7 weeks and 24 weeks after treatment commencement.
  Change in the the total score of Dysfunctional Beliefs and Attitudes about Sleep (DBAS-16)

CONTACTS AND LOCATIONS:
Overall Officials: RENATHA RAFIHI-FERREIRA, PHD, Principal Investigator — University of Sao Paulo General Hospital
Locations (1):
- University of Sao Paulo General Hospital., São Paulo, Brazil